CLINICAL TRIAL: NCT05703126
Title: Clinical and Diagnostic Significance of Endothelial Dysfunction and Myocardial Contractility in Patients With Acute Myeloid Leukemia
Brief Title: Clinical and Diagnostic Significance of Endothelial Dysfunction and Myocardial Contractility in Patients With AML
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samara State Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 77880421319552
Record Dates: First submitted 2022-12-19; First posted 2023-01-27 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Acute Myeloid Leukemia, Adult; Cardiotoxicity; Endothelial Dysfunction
Keywords: Acute Myeloid Leukemia; Cardiotoxicity; Endothelial Dysfunction; Polychemotherapy; Anthracyclines
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Cardiotoxicity | interventions — Medical History Taking; Anthropometry; Blood Cell Count; Echocardiography, Stress; Electrocardiography; Laser-Doppler Flowmetry

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The study group (Other): The study group will include patients with acute myeloid leukemia receiving chemotherapy, aged 18 to 65 years, without clinical signs of heart failure, with an LV ejection fraction of more than 50% before the start of polychemotherapy, in whom in the course of chemotherapy treatment after the next course of treatment a decrease in global longitudinal strain of 15% or more relative to the initial values will be revealed.
  Interventions: Diagnostic Test: History taking; Diagnostic Test: Anthropometry; Diagnostic Test: Complete blood count; Diagnostic Test: Biochemical blood test; Diagnostic Test: Coagulogram; Diagnostic Test: Immunoenzymatic analysis of the level of endothelin-1, asymmetric dimethylarginine; Diagnostic Test: Stress echocardiography with the definition of global longitudinal deformation of the myocardium; Diagnostic Test: Triplex scanning of neck vessels; Diagnostic Test: Electrocardiography; Diagnostic Test: Ultrasound of the abdominal cavity (with calculation of the area of the spleen) and lymph nodes; Diagnostic Test: Cytogenetic examination of the bone marrow to determine genetic abnormalities.; Diagnostic Test: Cytological examination of bone marrow cells with cytochemical examination; Diagnostic Test: Immunophenotypic examination of the bone marrow by flow cytometry; Diagnostic Test: Determination of the presence of a FLT3 mutation using the PCR Method; Diagnostic Test: laser Doppler flowmetry
- The control group (Other): The control group will consist of patients with acute myeloid leukemia receiving chemotherapy, aged 18 to 65 years, without clinical signs of heart failure, with an LV ejection fraction of more than 50% before the start of polychemotherapy, in whom no signs of myocardial disease will be detected during chemotherapy. and endothelial dysfunction.
  Interventions: Diagnostic Test: History taking; Diagnostic Test: Anthropometry; Diagnostic Test: Complete blood count; Diagnostic Test: Biochemical blood test; Diagnostic Test: Coagulogram; Diagnostic Test: Immunoenzymatic analysis of the level of endothelin-1, asymmetric dimethylarginine; Diagnostic Test: Stress echocardiography with the definition of global longitudinal deformation of the myocardium; Diagnostic Test: Triplex scanning of neck vessels; Diagnostic Test: Electrocardiography; Diagnostic Test: Ultrasound of the abdominal cavity (with calculation of the area of the spleen) and lymph nodes; Diagnostic Test: Cytogenetic examination of the bone marrow to determine genetic abnormalities.; Diagnostic Test: Cytological examination of bone marrow cells with cytochemical examination; Diagnostic Test: Immunophenotypic examination of the bone marrow by flow cytometry; Diagnostic Test: Determination of the presence of a FLT3 mutation using the PCR Method; Diagnostic Test: laser Doppler flowmetry

INTERVENTIONS:
Diagnostic Test: History taking — Careful history taking, including using questionnaires, to identify risk factors for the development of cardiovascular diseases using the SCORE scale.
Diagnostic Test: Anthropometry — Anthropometry: measurement of body weight and height. Calculation of body surface area using the Du Bois formula.
Diagnostic Test: Complete blood count — Before and after each course of chemotherapy: Complete blood count with counting the number of erythrocytes, leukocytes, leukocyte formula, platelets, erythrocyte sedimentation rate.
Diagnostic Test: Biochemical blood test — Before and after each course of chemotherapy: Biochemical blood test with the determination of the amount of total protein, total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides, creatinine, urea, AlAT, AsAT, LDH, glucose, C-reactive protein, troponin T, proBNP.
Diagnostic Test: Coagulogram — Before and after each course of chemotherapy: Coagulogram parameters (fibrinogen, APTT, INR).
Diagnostic Test: Immunoenzymatic analysis of the level of endothelin-1, asymmetric dimethylarginine — Before the start of the treatment and after each course of chemotherapy: Immunoenzymatic analysis of the level of endothelin-1, asymmetric dimethylarginine.
Diagnostic Test: Stress echocardiography with the definition of global longitudinal deformation of the myocardium — Before the start of the treatment and after each course of chemotherapy: Stress echocardiography with the definition of global longitudinal deformation of the myocardium.
Diagnostic Test: Triplex scanning of neck vessels — Before the start of the treatment and after each course of chemotherapy: Triplex scanning of neck vessels.
Diagnostic Test: Electrocardiography — Before and after each course of chemotherapy: Electrocardiography.
Diagnostic Test: Ultrasound of the abdominal cavity (with calculation of the area of the spleen) and lymph nodes — Before the start of the treatment and after each course of chemotherapy: Ultrasound of the abdominal cavity (with calculation of the area of the spleen) and lymph nodes.
Diagnostic Test: Cytogenetic examination of the bone marrow to determine genetic abnormalities. — Before the start of the treatment: Cytogenetic examination of the bone marrow to determine genetic abnormalities.
Diagnostic Test: Cytological examination of bone marrow cells with cytochemical examination — Before the start of the treatment and after each course of chemotherapy: Cytological examination of bone marrow cells with cytochemical examination.
Diagnostic Test: Immunophenotypic examination of the bone marrow by flow cytometry — Before the start of the treatment: Immunophenotypic examination of the bone marrow by flow cytometry.
Diagnostic Test: Determination of the presence of a FLT3 mutation using the PCR Method — Before the start of the treatment: Determination of the presence of a FLT3 mutation using the PCR Method.
Diagnostic Test: laser Doppler flowmetry — Before the start of the treatment and after each course of chemotherapy: Examination of microcirculation by laser Doppler flowmetry using the LAKK-OP apparatus (NPP Lazma, Moscow, 2011) with respiratory and occlusion tests.

SUMMARY:
Acute myeloid leukemia (AML) is a clonal neoplastic disease of the hematopoietic tissue associated with a mutation in the precursor cell of hematopoiesis, which results in a differentiation block and uncontrolled proliferation of immature myeloid cells.

Anthracycline antibiotics have been an integral part of the treatment of acute myeloid leukemia since the 1970s. However, the clinical usefulness of anthracyclines is limited primarily by the high incidence of cardiotoxicity. According to the European Society of Cardiology guidelines for cardio-oncology, cardiovascular toxicity is defined as any impairment of cardiac function associated with anticancer treatment, as the term encompasses both a wide range of possible clinical manifestations and an etiological relationship with various treatments, including chemotherapy, radiation therapy, immunotherapy and treatment with targeted drugs. Cardiovascular toxicity can be acute, subacute or delayed, manifesting many years after chemotherapy or radiation therapy, involving a number of cardiac structures, which can lead to the development of heart failure, coronary heart disease, valvular heart disease, arrhythmias, including cardiac conduction disorders and diseases of the pericardium.

Anthracycline-induced cardiotoxicity is the negative effect of anthracyclines on normal cardiac activity due to their toxic effects on the heart muscle and the cardiac conduction system. Anthracycline-induced cardiotoxicity manifests as asymptomatic left ventricular dysfunction in 57% of treated patients and restrictive or dilated cardiomyopathy leading to congestive heart failure (CHF) in 16% to 20% of patients. Anthracycline-induced congestive heart failure is often resistant to therapy and has a mortality rate of up to 79%. Thus, there is a need for early detection of cardiovascular dysfunction associated with chemotherapy treatment of acute myeloid leukemia in order to timely prescribe drug therapy.

Purpose of the study To optimize the early detection of endothelial dysfunction and left ventricular myocardial contractility in patients with acute myeloid leukemia during chemotherapy treatment based on a comprehensive assessment of instrumental and laboratory research parameters.

Expected results Based on a comprehensive analysis using laser Doppler flowmetry, stress echocardiography with the determination of global longitudinal strain of the myocardium, biochemical markers of endothelial damage and cardiac biomarkers, a correlation between violations of the contractility of the left ventricular myocardium and violations of the vasoregulatory function of the vascular endothelium will be revealed, which will allow developing an algorithm for early detection of cardiomyopathy and vascular complications in patients with acute myeloid leukemia during chemotherapy treatment.

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) is a clonal neoplastic disease of the hematopoietic tissue associated with a mutation in the precursor cell of hematopoiesis, which results in a differentiation block and uncontrolled proliferation of immature myeloid cells.

It is believed that AML affects an average of 3-5 people per 100,000 people per year. At the same time, the incidence increases sharply at the age of over 60 years and amounts to 12-13 cases per 100 thousand of the population in people over the age of 80 years. The median age of this disease is 65 years. With a population of 140 million inhabitants in Russia, the estimated incidence rate (according to European and American researchers) should be about 5 thousand cases.

Anthracycline antibiotics have been an integral part of the treatment of acute myeloid leukemia since the 1970s. Anthracycline is usually given for 3 days (eg, daunorubicin 45-90 mg/m 2 daily, idarubicin 12 mg/m 2 daily) in combination with cytarabine (100-200 mg/m 2 daily) continuously for 7 days ) ("7+3" mode). Anthracyclines block the synthesis of DNA and RNA by inhibiting the enzyme topoisomerase IIβ and mitochondrial topoisomerase I. The subsequent disruption of DNA replication and transcription prevents the proliferation of rapidly dividing cells. In addition, anthracyclines damage DNA, proteins, and cell membranes by creating free oxygen radicals.

The clinical usefulness of anthracyclines is limited primarily by the high incidence of cardiotoxicity. According to the European Society of Cardiology guidelines for cardio- oncology, cardiovascular toxicity is defined as any impairment of cardiac function associated with anticancer treatment, as the term encompasses both a wide range of possible clinical manifestations and an etiological relationship with various treatments, including chemotherapy, radiation therapy, immunotherapy and treatment with targeted drugs. Cardiovascular toxicity can be acute, subacute or delayed, manifesting many years after chemotherapy or radiation therapy, involving a number of cardiac structures, which can lead to the development of heart failure, coronary heart disease, valvular heart disease, arrhythmias, including cardiac conduction disorders, and diseases of the pericardium.

Anthracycline-induced cardiotoxicity is the negative effect of anthracyclines on normal cardiac activity due to their toxic effects on the heart muscle and the cardiac conduction system. It is believed to be mediated in part by reactive oxygen species generated by anthracycline treatment, which leads to lipid peroxidation and DNA damage in cardiomyocytes. Other putative causes of anthracycline-induced cardiotoxicity include accumulation of cardiotoxic anthracycline metabolites in the heart, disruption of calcium homeostasis, mitochondrial damage, and induction of apoptosis.

Anthracycline-induced cardiotoxicity manifests as asymptomatic left ventricular dysfunction in 57% of treated patients and restrictive or dilated cardiomyopathy leading to congestive heart failure (CHF) in 16% to 20% of patients. Anthracycline-induced congestive heart failure is often resistant to therapy and has a mortality rate of up to 79%. Thus, there is a need for early detection of cardiovascular dysfunction associated with chemotherapy treatment of acute myeloid leukemia in order to timely prescribe drug therapy.

Purpose of the study To optimize the early detection of endothelial dysfunction and left ventricular myocardial contractility in patients with acute myeloid leukemia during chemotherapy treatment based on a comprehensive assessment of instrumental and laboratory research parameters.

Research objectives

1. To assess the state of endothelial function in patients with acute myeloid leukemia receiving chemotherapy based on a comprehensive assessment, including laser Doppler flowmetry and biochemical markers of endothelial damage (endothelin-1, asymmetric dimethylarginine).
2. To characterize the contractility of the left ventricular myocardium in patients with acute myeloid leukemia during chemotherapeutic treatment based on the indicators of stress echocardiography with the determination of global longitudinal deformation of the myocardium, as well as to assess the presence of myocardial damage by determining the level of highly sensitive troponin and brain natriuretic peptide.
3. To study the relationship between dynamic indicators of microcirculation, determined by laser Doppler flowmetry, with indicators of contractility of the left ventricular myocardium, detected using stress echocardiography with the determination of global longitudinal deformation of the myocardium, and the results of laboratory methods for assessing the function of the endothelium and myocardium.
4. To determine the frequency of development of various phenotypes of cardiovascular toxicity.
5. To identify the most significant prognostic criteria for the development of cardiotoxicity in patients with acute myeloid leukemia receiving chemotherapy.

Scientific novelty

1. For the first time, an algorithm for early detection of endothelial dysfunction and left ventricular myocardial contractility in patients with acute myeloid leukemia during chemotherapy treatment will be developed.
2. For the first time, the vasoregulatory function of the endothelium and the contractility of the left ventricular myocardium in patients with acute myeloid leukemia receiving chemotherapy will be studied based on a comprehensive assessment using laser Doppler flowmetry, stress echocardiography with the determination of global longitudinal deformation of the myocardium, biochemical markers of endothelial damage and cardiac biomarkers.

Practical significance It is planned to develop an algorithm for early detection of endothelial dysfunction and left ventricular myocardial contractility in patients with acute myeloid leukemia during chemotherapy treatment based on a comprehensive assessment using laser Doppler flowmetry, stress echocardiography with the determination of global longitudinal myocardial strain, biochemical markers of endothelial damage and cardiac biomarkers. .

Expected results Based on a comprehensive analysis using laser Doppler flowmetry, stress echocardiography with the determination of global longitudinal strain of the myocardium, biochemical markers of endothelial damage and cardiac biomarkers, a correlation between violations of the contractility of the left ventricular myocardium and violations of the vasoregulatory function of the vascular endothelium will be revealed, which will allow developing an algorithm for early detection of cardiomyopathy and vascular complications in patients with acute myeloid leukemia during chemotherapy treatment.

Research hypothesis:

The proposed algorithm for the early detection of cardiovascular complications in patients with acute myeloid leukemia receiving chemotherapy treatment is an effective method for diagnosing cardiovascular complications at subclinical stages for the timely initiation of their therapy.

Study Design In total, it is planned to study 100 patients with acute myeloid leukemia receiving chemotherapy, aged 18 to 65 years, without clinical signs of heart failure, with an LV ejection fraction of more than 50% before the start of polychemotherapy.

The study group will include patients with acute myeloid leukemia receiving chemotherapy, aged 18 to 65 years, without clinical signs of heart failure, with an LV ejection fraction of more than 50% before the start of polychemotherapy, in whom in the course of chemotherapy treatment after the next course of treatment a decrease in global longitudinal strain of 15% or more relative to the initial values will be revealed.

The control group will consist of patients with acute myeloid leukemia receiving chemotherapy, aged 18 to 65 years, without clinical signs of heart failure, with an LV ejection fraction of more than 50% before the start of polychemotherapy, in whom no signs of myocardial disease and endothelial dysfunction will be detected during chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* patients with acute myeloid leukemia receiving anthracycline-containing polychemotherapy regimens aged 18 to 65 years, without clinical signs of heart failure, with an LV ejection fraction of more than 50% before starting chemotherapy;
* availability of informed consent of the patient to participate in the study.

Exclusion Criteria:

* acute violation of cerebral circulation in history;
* a history of myocardial infarction;
* the presence of diabetes mellitus type I and II;
* the presence of chronic kidney disease C1-C5 stages;
* the presence of stable angina III-IV functional classes;
* the presence of unstable angina pectoris;
* the presence of atrial fibrillation and flutter;
* the presence of arterial hypertension of 2-3 degrees;
* the presence of other oncological diseases;
* inflammatory diseases in the acute stage;
* diseases of the thyroid gland;
* therapy with any monoclonal antibodies in history;
* a positive test for the presence of HIV and hepatitis B and C;
* alcoholism, drug addiction;
* the presence of neuroleukemia, extramedullary foci of leukemia;
* refusal of the patient to be examined.
* the emergence of life-threatening situations during the study;
* development in patients of diseases related to the non-inclusion criteria;
* refusal of the patient to further examination.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-08-03 (Estimated)

PRIMARY OUTCOMES:
Change of global longitudinal strain of 15% or more relative to the initial values | Evaluation is carried out within 1 week after each course of chemotherapy up to 10 months, evaluated after each course of induction of remission and consolidation of remission.
  Change of global longitudinal strain of the myocardium according to stress echocardiography by 15% or more relative to the values obtained before the start of chemotherapy treatment.

SECONDARY OUTCOMES:
Change of the index of microcirculation according to laser Doppler flowmetry | Evaluation is carried out within 1 week after each course of chemotherapy up to 10 months, evaluated after each course of induction of remission and consolidation of remission.
  Change of the microcirculation index according to the results of laser Doppler flowmetry in relation to the values obtained before the start of chemotherapy treatment.
Change of the Coefficient of Variation of Microcirculation According to Laser Doppler Fluometry | Evaluation is carried out within 1 week after each course of chemotherapy up to 10 months, evaluated after each course of induction of remission and consolidation of remission.
  Change of the coefficient of variation of microcirculation according to the results of laser Doppler flowmetry in relation to the values obtained before the start of chemotherapy treatment.
Change of the level of highly sensitive T-troponin | Evaluation is carried out within 1 week after each course of chemotherapy up to 10 months, evaluated after each course of induction of remission and consolidation of remission.
  Change of the level of highly sensitive T-troponin, which goes beyond the reference values, in relation to the values obtained before the start of chemotherapy treatment.
Change of brain natriuretic peptide level | Evaluation is carried out within 1 week after each course of chemotherapy up to 10 months, evaluated after each course of induction of remission and consolidation of remission.
  Change of the level of brain natriuretic peptide that goes beyond the reference values, in relation to the values obtained before the start of chemotherapy treatment.
Change of the level of asymmetric dimethylarginine | Evaluation is carried out within 1 week after each course of chemotherapy up to 10 months, evaluated after each course of induction of remission and consolidation of remission.
  Change of the level of asymmetric dimethylarginine that goes beyond the reference values, in relation to the values obtained before the start of chemotherapy treatment.
Change of the level of endothelin-1 | Evaluation is carried out within 1 week after each course of chemotherapy up to 10 months, evaluated after each course of induction of remission and consolidation of remission.
  Change of the level of endothelin-1, which goes beyond the reference values, in relation to the values obtained before the start of chemotherapy treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Igor Davydkin, Principal Investigator — Samara State Medical University
Locations (1):
- Clinics of the Samara Medical University, Samara, Samara Oblast, Russia

IPD SHARING:
Plan to Share IPD: Undecided